CLINICAL TRIAL: NCT03410186
Title: Effectiveness of a Continuous Paravertebral Analgesia Via Erector Spinae Plane (ESP) Catheters Within a Strict Enhanced Recovery Protocol (ERP) in Adult Patients Following Open Radical Cystectomy (ORC): an Observational Pilot Study
Brief Title: Effectiveness of Continuous Erector Spinae Plane and Intrathecal Opioid (ESPITO) Analgesia in Open Radical Cystectomy
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE102914
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Open Radical Cystectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Bowel dysfunction is a major complication following open surgery for invasive cancer of the bladder that causes significant discomfort, complications and prolongs the length of stay in the hospital. Amenable factors that are responsible for postoperative bowel dysfunction include intravenous morphine given for pain relief and epidural infusion requiring excess intravenous fluids administration after surgery. The British Association of Urological Surgeons (BAUS) have published the Enhanced Recovery protocol (ERP) to reduce length of hospital stay following open surgery for cancer of the urinary bladder. The ERP is a care package that is provided to the patient from the day of the surgery till hospital discharge. At Leicester, we have modified the ERP and this has become the standard of care for our patients undergoing this surgery. The modified ERP care package includes a novel combination of two established pain relief techniques (erector spinae plane analgesia and intrathecal opioids) that will avoid the use of epidural analgesia, excess intravenous fluids administration and intravenous morphine in the postoperative period. The modified ERP has been well accepted by the patients and the clinical team looking after these patients. We would like to perform a formal evaluation of the modified ERP care package in the management of adult patients undergoing open bladder surgery through an observational pilot study.

Aim of the study is to evaluate the incidence of postoperative bowel dysfunction and the median length of hospital stay in adult patients undergoing(open radical cystectomy Methods: Prospective, observational pilot study that will be conducted at Leicester General Hospital over 24 months. Adult patients scheduled to undergo open radical cystectomy will be included in the study. Patients who will have laparoscopic surgery will be excluded. After providing written consent, the participants will receive an enhanced recovery protocol (ERP) care package that will commence from the day of their surgery till they are discharged from the hospital. Participants will be asked to report time of opening their bowel, pain scores on movement, presence of nausea and vomiting, bowel dysfunction, length of hospital stay and any complication from day of surgery till 30 days after surgery. Participation in the study will end at 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients scheduled to undergo open radical cystectomy
2. American Society of Anesthesiologists (ASA) 2 or 3

Exclusion Criteria:

1. Lack of consent including from those participants who lack mental capacity to give informed consent
2. American Society of Anesthesiologists (ASA) 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is based on a cohort of adult patients scheduled to undergo elective open radical cystectomy for muscle invasive carcinoma of the urinary bladder.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
The incidence of Post Operative Ileus (POI) | 24 months
  The incidence of postoperative ileus (POI): POI is defined as 'Intolerance of solid food at the 5th postoperative day with the need to hold oral nutrition because of bloating, nausea and vomiting'

SECONDARY OUTCOMES:
The length of hospital stay | 24 months
  Defined as duration from the day of surgery to the day the participant meets the following 4 criteria: Pain Free, Ambulant, Bowels Opened & Stoma Trained

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided